CLINICAL TRIAL: NCT04132973
Title: An Acceptability and Feasibility Study of a Compassion-Based Guided Self-Help Intervention for Depression in People With Skin Conditions.
Brief Title: Investigating Compassion-Based Guided Self-Help for Depression in People With Skin Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 163781
Record Dates: First submitted 2019-10-17; First posted 2019-10-21 (Actual); Results first posted 2021-10-26 (Actual); Last update posted 2021-10-26 (Actual); Status verified 2019-10

CONDITIONS: Dermatologic Disease; Depression
Keywords: acceptability; feasibility; self-management
MeSH Terms: conditions — Skin Diseases; Depression

STUDY DESIGN:
Intervention Model Description: This is an acceptability and feasibility study of a novel healthcare intervention, therefore there is only one study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compassion guided self-help (Experimental): Participants will engage in a six-week online compassion-based self-help programme with email guidance from the researcher.
  Interventions: Behavioral: Compassion for Skin Conditions

INTERVENTIONS:
Behavioral: Compassion for Skin Conditions — Online guided self-help intervention derived from Compassion Focused Therapy (Gilbert, 2010).

SUMMARY:
The study aims to explore whether an online compassion-based guided self-help intervention is perceived as acceptable to people with heterogeneous skin conditions, in terms of retention rates and explicit feedback. The study also aims to investigate the feasibility of providing online compassion-based self-help and email guidance. Changes in depression, self-compassion and skin-related distress will be assessed to give an estimate of likely effect sizes for future research

DETAILED DESCRIPTION:
The study will investigate an online compassion-based self-help intervention with email guidance with people with skin conditions who are experiencing depressive symptoms. As the study aims to investigate a novel intervention, the study will be an acceptability and feasibility study that uses a pre-post design. Participants with skin conditions will be recruited from the general population using online methods (social media and advertisements on skin condition charities/organisations websites). Participants will complete baseline measures using Qualtrics and then be able to commence a six-week online intervention, consisting of a dedicated website containing six self-help sessions to work through. Regular guidance will be provided by the researcher via email. The self-help exercises in the current study will consist of a number of exercises derived from Compassion Focused Therapy (CFT)/Compassionate Mind Training, such as using soothing rhythm breathing, compassionate imagery and compassionate writing. Explicit feedback will be sought from participants at the end of each session, and at the end of the intervention overall. Engagement with the website will be monitored via user logins and this will be used to calculate the retention rate for the intervention. Post-intervention measures will be collected one week after the end of the intervention. All participants will be provided with signposting information relating to mental health and skin conditions, and advised to see their GP if they require any further support with their physical or mental health.

Intervention The guided self-help intervention will consist of six online sessions of self-help information for participants to work through, plus activities to carry out in-between sessions. The intervention will consist of psycho-education material, self-monitoring, and compassion-inducing exercises from CFT. The self-help exercises in the intervention will be evidence-based as being effective for depression: the compassion-focused imagery exercises and the letter-writing exercise will be based on those used in published studies. Other exercises, such as thought monitoring and relapse prevention planning, are commonly used in cognitive behavioural therapy (CBT) and, as CFT is an adapted form of CBT, will be included in the current self-help intervention. The session content and homework exercises will build on previous sessions and homework, so there will be a clear sense of progression through the intervention. In addition, imagery and written homework exercises will be alternated, to provide variety and keep participants engaged in the intervention. Examples relating to skin conditions will be given throughout the self-help materials. Expert feedback regarding the content of the website has been sourced through personal contacts and social media. Feedback has already been gathered from three people with skin conditions. Changes to the website deemed necessary based on their feedback have been made.

Data analysis strategy Text responses from participants' feedback on the intervention overall will be analysed using content analysis to identify helpful aspects of the intervention and areas for improvement. Quantitative data (outcome measures and acceptability ratings) will be screened for outliers and missing values, and descriptive statistics will be conducted for all variables. The data will be tested for the assumption of normality. Paired t-tests will be used to test for differences in participants' psychological outcome measures before and after the intervention. This information will also be used to calculate effect sizes (dz) for changes in scores on each outcome measure. Intention-to-treat and completer analyses will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* self-report of currently having a skin condition that has been present for at least the last six months and has been diagnosed by a medical professional.
* scored 10-20 (inclusive) on DASS-DEP (depression subscale of Depression Anxiety Stress Scales).

Exclusion Criteria:

* currently receiving a psychological therapy for a mental health problem.
* current diagnosis of a serious mental illness (e.g. psychosis or bipolar disorder).
* current diagnosis of a drug or alcohol problem.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-04-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Elaine N Clarke, PhD, Principal Investigator — University of Sheffield
Locations (1):
- The University of Sheffield, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Individual patient data will not be made available to maintain confidentiality, but aggregated data may be made available from the lead researcher upon reasonable request.

REFERENCES:
- [Background] Kelly AC, Zuroff DC, Shapira LB. Soothing oneself and resisting self-attacks: The treatment of two intrapersonal deficits in depression vulnerability. Cognitive Therapy and Research 33: 301-313, 2009.
- [Background] Shapira LB, Mongrain M. The benefits of self-compassion and optimism exercises for individuals vulnerable to depression. The Journal of Positive Psychology 5: 337-389, 2010.
- [Background] McEwan K, Gilbert P. A pilot feasibility study exploring the practising of compassionate imagery exercises in a nonclinical population. Psychol Psychother. 2016 Jun;89(2):239-43. doi: 10.1111/papt.12078. Epub 2015 Oct 10. PMID 26454144
- [Background] Gilbert P, Irons C. Focused therapies and compassionate mind training for shame and self-attacking. In: Gilbert P, editor. Compassion: Conceptualisations, Research and Use in Psychotherapy. Hove: Routledge; 2005. p 263-325.
- [Background] Gilbert P. Compassion Focused Therapy: The CBT distinctive features series. Hove: Routledge; 2010. 237 p.
- [Derived] Clarke EN, Norman P, Thompson AR. Online compassion-based self-help for depression in people with skin conditions: a feasibility study. Pilot Feasibility Stud. 2024 Apr 16;10(1):63. doi: 10.1186/s40814-024-01486-4. PMID 38627850

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Compassion Guided Self-help
Started | 34
Completed Intervention | 11
Completed | 8
Not Completed | 26

BASELINE CHARACTERISTICS:
Arm/Group | Compassion Guided Self-help
Number analyzed (Participants) | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.2 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 3
Race/Ethnicity, Customized [Number; unit: participants]
  White | 28
  British Pakistani | 1
  British African | 1
  Mixed heritage | 2
  Japanese | 1
  Not specified | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 31
  Italy | 1
  Malaysia | 1
  Spain | 1
Skin condition (self-reported) [Number; unit: participants]
  Eczema | 16
  Psoriasis | 13
  Other | 11

OUTCOME MEASURES:

1. Primary Outcome: Acceptability of Intervention Overall
Description: Percentage of participants that log in to the online intervention during their sixth week (i.e. participant retention).
Time Frame: Week 6 for each participant (rolling recruitment).
Measure: Count of Participants; unit: Participants
Arm/Group | Compassion Guided Self-help
Number analyzed (Participants) | 34
Participants | 11

2. Primary Outcome: Acceptability of Session 1
Description: Likert scale ratings for acceptability components (ease of use, helpfulness of information, ease of understanding, adequacy of information, and visual appeal) for each weekly session. These items have been adapted from the Website Evaluation Questionnaire as no suitable validated measure could be found. Scale mean scores range from 0 to 4, with higher scores indicating higher perceived acceptability.
Time Frame: Day 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compassion Guided Self-help
Number analyzed (Participants) | 16
score on a scale | 2.35 (1.28)

3. Primary Outcome: Acceptability of Session 2
Description: as for outcome 2
Time Frame: Day 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compassion Guided Self-help
Number analyzed (Participants) | 13
score on a scale | 2.35 (1.30)

4. Primary Outcome: Acceptability of Session 3
Description: as for outcome 2
Time Frame: Day 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compassion Guided Self-help
Number analyzed (Participants) | 9
score on a scale | 2.56 (1.13)

5. Primary Outcome: Acceptability of Session 4
Description: as for outcome 2
Time Frame: Day 22
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compassion Guided Self-help
Number analyzed (Participants) | 5
score on a scale | 2.7 (1.29)

6. Primary Outcome: Acceptability of Session 5
Description: as for outcome 2
Time Frame: Day 29
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compassion Guided Self-help
Number analyzed (Participants) | 7
score on a scale | 2.43 (1.36)

7. Primary Outcome: Acceptability of Session 6
Description: as for outcome 2
Time Frame: Day 36
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compassion Guided Self-help
Number analyzed (Participants) | 5
score on a scale | 2.97 (1.25)

8. Secondary Outcome: Change From Baseline Depression Subscale of the Depression Anxiety Stress Scales (DASS-DEP) Score After Six Weeks.
Description: Self-report measure of depression. Measure ranges from 0 to 42, with higher scores indicating higher levels of depressive symptomatology.
Time Frame: Days 1 and 43.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compassion Guided Self-help
Number analyzed (Participants) | 8
score on a scale | -7.75 (7.03)

9. Secondary Outcome: Change From Baseline Self-Compassion Scale (SCS) Score After Six Weeks.
Description: Self-report measure of self-compassion. Measure ranges from 26 to 130, with higher scores indicating higher levels of self-compassion.
Time Frame: Days 1 and 43.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compassion Guided Self-help
Number analyzed (Participants) | 8
score on a scale | 17.88 (27.82)

10. Secondary Outcome: Change From Baseline Dermatology Life Quality Index (DLQI) Score After Six Weeks.
Description: Self-report measure of impact of skin condition on quality of life. Measure ranges from 0 to 30, with higher scores indicating higher effect of the skin condition on the person's life.
Time Frame: Days 1 and 43.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Compassion Guided Self-help
Number analyzed (Participants) | 8
score on a scale | -6.38 (6.61)

ADVERSE EVENTS:
Time Frame: Rolling recruitment: from baseline for each participant until data collection ended on Day 42. Participants also were able to contact the lead researcher by email after this point (no fixed end point for this).
Arm/Group | Compassion Guided Self-help
All-Cause Mortality (participants affected / at risk) | 0/34
Serious Adverse Events (participants affected / at risk) | 0/34
Other Adverse Events (participants affected / at risk) | 3/34
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Compassion Guided Self-help (N=34)
Psychological distress (Psychiatric disorders) | 3 (3) — Any psychological distress, however minor, experienced as a result of taking part in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-09): https://cdn.clinicaltrials.gov/large-docs/73/NCT04132973/Prot_SAP_000.pdf
  • Informed Consent Form (2019-11-15): https://cdn.clinicaltrials.gov/large-docs/73/NCT04132973/ICF_001.pdf